CLINICAL TRIAL: NCT00858910
Title: Comparison of Embedded and Added Motor Imagery Training to Improve a Motor Skill in Patients After Stroke: a Pilot Randomised Controlled Trial Using a Mixed Methods Approach
Brief Title: Comparison of Embedded and Added Motor Imagery Training in Patients After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reha Rheinfelden (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Prof. Thierry Ettlin, Reha Rheinfelden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/077
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2010-07

CONDITIONS: Stroke
Keywords: Motor imagery; Motor skill; Performance improvement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EG1: embedded MI (Experimental): Experimental group 1:
  Participants receive motor imagery (MI) training included in 45min physiotherapy, 3 times per week for 2 weeks.
  Interventions: Other: Motor imagery (MI) training
- EG2: added MI (Experimental): Experimental group 2:
  Participants receive a 15 minutes motor imagery (MI) training added to a 30 min physiotherapy session, 3 times a week for two weeks.
  Interventions: Other: Motor imagery (MI) training
- CG (Placebo Comparator): Control group:
  Participants receive a 15 min control intervention added to their 30 min physiotherapy session, 3 times a week for two weeks.
  Interventions: Other: Control intervention

INTERVENTIONS:
Other: Motor imagery (MI) training — MI training encloses the internal rehearsal of a known motor skill without any overt motor output.
  Arms: EG1: embedded MI; EG2: added MI
Other: Control intervention — The control intervention encloses relaxation and breathing exercises, and information about:
  * the disease (stroke),
  * therapy options,
  * self-help groups and their offers for support,
  * helping aids for independent living at home.
  Arms: CG

SUMMARY:
The purpose of the study is to examine if patients in the embedded motor imagery (MI) training group (EG1) need less time to perform the motor task than patients in the added MI training group (EG2).

DETAILED DESCRIPTION:
The purpose of the study is to examine if patients in the embedded MI training into physiotherapy (EG1) need less time to perform the motor task than patients in the added MI training to physiotherapy (EG2).

A third groups serves a control group (CG) to investigate the effect of the intervention versus a group with a control intervention.

Additionally, semi-structured interviews before and after the intervention will give an insight in the patient's experience with motor imagery (MI), their expectations regarding the intervention and their opinions about MI after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients after a first-ever ischemic or hemorrhagic stroke
* Outpatients or leaving inpatients 3 months after stroke
* Ability to stand with or without a cane for at least 30 sec on a normal hard floor
* Ability to walk for 20 metres with or without a cane or an orthosis
* MMSE with at least 20 points
* Age older than 18 years
* Signed written informed consent

Exclusion Criteria:

* Joint replacements (knee, hip, shoulder)
* Limiting pain in the upper or lower body
* Limiting range of motion (ROM) in the hip, knee, ankle joint or toes
* Body weight more than 90 kilograms
* Compromised mental capacity to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Time in seconds to perform a motor task: "Going down, laying on the floor and getting up again." | 2 weeks

SECONDARY OUTCOMES:
Further outcome measures: - Help needed to perform the task, scored on a 7-item scale (1 total help, 7 completely independent) - Stage of motor task (one out of 13 possible stages) | 2 weeks
Motor impairment and independence measured with the extended Barthel index (EBI). | 2 weeks
Balance measured with the Berg Balance Scale (BBS). | 2 weeks
Motor imagery ability measured with the kinesthetic and visual motor imagery questionnaire (KVIQ) and the 'Imaprax 1.1' software. | 2 weeks
Fear of falling (FOF) is measured with the Activities-Specific Balance Confidence Scale (ABC-scale). | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation centre: Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Zimmermann-Schlatter A, Schuster C, Puhan MA, Siekierka E, Steurer J. Efficacy of motor imagery in post-stroke rehabilitation: a systematic review. J Neuroeng Rehabil. 2008 Mar 14;5:8. doi: 10.1186/1743-0003-5-8. PMID 18341687
- [Derived] Schuster C, Butler J, Andrews B, Kischka U, Ettlin T. Comparison of embedded and added motor imagery training in patients after stroke: results of a randomised controlled pilot trial. Trials. 2012 Jan 23;13:11. doi: 10.1186/1745-6215-13-11. PMID 22269834
- [Derived] Schuster C, Butler J, Andrews B, Kischka U, Ettlin T. Comparison of embedded and added motor imagery training in patients after stroke: study protocol of a randomised controlled pilot trial using a mixed methods approach. Trials. 2009 Oct 22;10:97. doi: 10.1186/1745-6215-10-97. PMID 19849835